CLINICAL TRIAL: NCT01284712
Title: Natural Killer Cells and Polycythemia Vera (Vaquez's Disease)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/16; 2009-A00395-52
Record Dates: First submitted 2009-08-03; First posted 2011-01-27 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Polycythemia Vera
Keywords: treatment by bleedings
MeSH Terms: conditions — Polycythemia Vera | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood sample — blood sample coming from therapeutic bleeding in hospital

SUMMARY:
Natural Killer cells (NK) are pivotal cells of innate immunity, that sense defective expression of HLA class I molecules and are complementary to specific cytotoxic T lymphocytes. A defect in NK cell cytotoxicity has been described in some hematopoietic malignancies such as acute myeloid leukemia, multiple myeloma, myelodysplastic syndroms. This defect is at least partially linked to a decreased or absent expression of some activating NK cell molecules, more particularly the so-called Natural Cytotoxicity Receptors (NCRs) NKp30, NKp44 and NKp46. Some old publications have demonstrated defective NK cytotoxicity in myeloproliferative syndroms (chronic myeloid leukemia, primary thrombocytosis, polycythemia vera). The investigators more particularly focused their attention on polycythemia vera (Vaquez's disease), a myeloproliferative disease characterized by the recently describet mutation V617F of the JAK2 tyrosine kinase. The investigators will precise the mechanisms leading to this cytotoxicity defect, the investigators also will evaluate the implication of V617F mutation on NK physiology, and will study the interactions between NK cells and hematopoietic progenitors.

ELIGIBILITY:
Inclusion Criteria:

* Polycythemia vera
* Treatment by therapeutic bleedings
* No cytotoxic treatment during the previous six months

Exclusion Criteria:

* No Polycythemia vera
* No treatment by therapeutic bleedings
* Cytotoxic treatment during the previous six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VAQUEZ'S DISEASE
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To describe immunologic anomalies in polycythemia vera | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Regis Costello, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France